CLINICAL TRIAL: NCT06145451
Title: Caregiver Relational Responsiveness (RR): An Understudied Fidelity Construct as a Mechanism to Increase Protective Factors Against Maltreatment
Brief Title: Connected Through Coaching for Flourishing Families
Acronym: CCFF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Ohio State University (Other); Case Western Reserve University (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Deborah Moon, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY23110074; 1 K01CE003543-01-00 (Other Grant/Funding Number: Centers for Disease Control and Prevention); 1K01CE003543-01 (NIH)
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Maltreatment by Parent
Keywords: maltreatment prevention, relational responsiveness

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Researchers have no direct contact with research participants as all data collection activities are carried out by care providers.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): The Family Success Network is a multi-tier, multi-component community-based maltreatment prevention program that offers tailored preventive services for caregivers of children aged 0-18. Average lengths of service completion is approximately 3 months.
  Interventions: Behavioral: Family Success Network
- Waitlist Control Group (No Intervention): Families in the Control Group will not receive any FSN services except concrete support of upto $500.

INTERVENTIONS:
Behavioral: Family Success Network — The Family Success Network (FSN) is a community-based maltreatment prevention program that is being piloted to serve caregivers of children aged between 0-18 in the Trumbull, Mahoning, and Columbiana Counties in Ohio. FSN is a comprehensive multi-tier program providing information and referrals to community resources at Tier I (i.e., the initial contact stage), caregiver education, and financial literacy program along with concrete support at Tier II (i.e., enrollment in family coaching services in FSN), and a life skills program and monthly home visits for families with more intensive needs at tier III (most intensive level of FSN services).
  Other Names: FSN
  Arms: Treatment group

SUMMARY:
Despite the known association between the quality of participant relational engagement with service providers and clinical outcomes, limited studies have examined caregiver Relational Responsiveness (RR) as a mechanism to achieve maltreatment prevention program outcomes. Using a realist-informed mixed method approach, this study will examine RR's role in mediating the effects of a community-based maltreatment prevention program, the Family Success Network (FSN) on protective factors against maltreatment and the contexts within which RR's mediation effects are activated or inhibited.

DETAILED DESCRIPTION:
Maltreatment prevention programs can promote public health by building protective factors among at-risk families. To maximize their benefits, programs should be delivered as intended by maintaining fidelity. Participant responsiveness (PR) is an under-studied fidelity construct defined as the degree to which participants "respond to or are engaged by" intervention at the behavioral, attitudinal, and relational levels. However, previous studies mostly focus on behavioral and attitudinal responsiveness such as attendance, follow-through, and satisfaction. The purpose of this study is to examine the role of participant Relational Responsiveness (RR) as a mechanism to increase protective factors against child maltreatment among the caregivers participating in the Family Success Network (FSN). The FSN is a community-based maltreatment prevention program piloted to serve 3 under-served counties in Ohio with high maltreatment rates. In FSN, coaches and families collaboratively develop a tailored plan of services designed to increase family protective factors. Focusing on primary and secondary prevention, FSN serves families with no history of substantiated maltreatment. Leveraging the parent study (clinicatrials registration currently in progress), which is a Randomized Controlled Trial (RCT) funded by the Children's Bureau, the proposed study will pursue the following aims; 1) To examine the structural validity of the Relational Responsiveness (RR) measure among FSN participants; 2) To determine the degree to which RR mediates FSN effects and whether RR's mediation effects are moderated by caregiver race and gender; 3) To identify contexts within which RR's mediation effects are activated or inhibited using a realist informed mixed-method approach. The parent study focuses on FSN outcome and process evaluations. Aims 1 and 2 of this study will utilize quantitative data collected through the parent RCT (protective factors and Working Alliance Inventory-Short Revised). Aim 3 will use mixed data involving the quantitative data collected through the parent RCT and the qualitative data to be collected in this study.

ELIGIBILITY:
Inclusion Criteria:

* Being an adult primary caregiver living in the tri-county area
* Having at least one child aged between 0-17
* Reporting at least one maltreatment risk factor at the time of intake
* Receiving family coaching services at Tier II and above in FSN.

Exclusion Criteria:

* Having a substantiated history of child maltreatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 612 (Estimated)
Dates: Start 2024-08-16 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Protective factors | baseline vs. 3 month (at the time of service completion)
  The family protective factors will be assessed using the Protective Factors Survey - Second Edition (PFS-2). It is a 19-item, 5-point Likert scale assessing 1) Family Functioning/Resilience [family's adaptive skills and strategies to persevere in times of crisis, 3 items, subscale score of 0-3], 2) Nurturing/Attachment [emotional bond and positive parent-child interactions, 4 items, subscale score of 0-4]; 3) Concrete Supports [perceived access to tangible goods and services, 2 items, subscale score of 0-8]; 4) Social Supports [4 items, subscale score of 0-16 plus the number of items checked in the social support checklist, which ranges between 0-4]. Except for the concrete support subscale in which higher scores indicate lower level of concrete support, higher scores indicate higher level of assessed qualities in all the other subscales.

SECONDARY OUTCOMES:
Relational Responsiveness | baseline vs. 3 month (at the time of service completion)
  Participant relational responsiveness (RR) will be assessed using the Working Alliance Inventory Short-Revised (WAI-SR), which is a 12-item, 5-point Likert scale with the response categories ranging from "Seldom" to "Always". WAI consists of three domains including agreement on goals, agreement on tasks, and bond between clients and providers. Instead of aggregating multiple items into a continuous variable, RR will be treated as a single order continuous latent construct with 3 distinct domains.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Moon, PhD, Principal Investigator — University of Pittsburgh
Locations (3):
- United States (3):
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
De-identified qualitative data may be shared upon request.

REFERENCES:
- [Background] Collaborative fidelity assessment planning for the evaluation of a community-based maltreatment prevention model: The family success network (FSN) D. J. Moon, M. Johnson-Motoyama, C. Bailey Nichols, N. Rolock, H. Haran and R. Bai Children and Youth Services Review 2022 Vol. 137 Pages 106457 DOI: https://doi.org/10.1016/j.childyouth.2022.106457
- [Background] Johnson-Motoyama M, Moon D, Rolock N, Crampton D, Nichols CB, Haran H, Zhang Y, Motoyama Y, Gonzalez E, Sillaman N. Social Determinants of Health and Child Maltreatment Prevention: The Family Success Network Pilot. Int J Environ Res Public Health. 2022 Nov 21;19(22):15386. doi: 10.3390/ijerph192215386. PMID 36430105